CLINICAL TRIAL: NCT00430547
Title: Thyroid-Associated Ophthalmopathy Subtypes and Orbital Antibodies
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Barwon Health (Other Government)
Collaborators: University of Melbourne (Other); National Health and Medical Research Council, Australia (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 03/53
Record Dates: First submitted 2007-02-01; First posted 2007-02-02 (Estimated); Last update posted 2007-02-02 (Estimated); Status verified 2003-08

CONDITIONS: Graves' Ophthalmopathy
MeSH Terms: conditions — Graves Ophthalmopathy | interventions — Carbimazole; Iodine-131

INTERVENTIONS:
Drug: Carbimazole, radio-active iodine (I131)

SUMMARY:
The purpose of this study is to determine whether radioactive iodine, as compared to anti-thyroid medications, is a risk factor for the development or progression of thyroid-associated ophthalmopathy in patients with hyperthyroidism due to Graves' disease. The other aim of this study is to determine the incidence of the various ophthalmopathy subtypes and the utility of orbital antibodies in the diagnosis, classification and monitoring of patients with thyroid-associated ophthalmopathy.

ELIGIBILITY:
Inclusion Criteria:

* Graves' disease diagnosed in the last 3 months, regardless of the presence of ophthalmopathy

Exclusion Criteria:

* Pre-existing eye disease: e.g. orbital surgery, orbital irradiation or significant loss of vision
* Age < 18 years
* Inability to consent to participation in the study
* Pregnancy
* History of radio-active iodine therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60
Dates: Start 2003-08; Study Completion 2006-01

PRIMARY OUTCOMES:
Onset or progression of ophthalmopathy following radio-active iodine therapy

CONTACTS AND LOCATIONS:
Overall Officials: Jack R Wall, BMBS, FRACP, PhD, Principal Investigator — University of Sydney
Locations (1):
- Barwon Health - The Geelong Hospital, Geelong, Victoria, Australia